CLINICAL TRIAL: NCT04146727
Title: Utilizing Technology for Optimization of Pain Management and Mobilization in High Risk Cardiac Surgical ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Anahat Dhillon, Staff Physician II, Cedars-Sinai Medical Center
Other Study IDs: pro000578722
Record Dates: First submitted 2019-10-24; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Transplant; Failure, Heart; Heart Failure, Congestive; Lung Transplant Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICU Duration: The total study duration is determined by their length of stay in the ICU.
- Transplant through 1 month at Home: Time from surgery through 1 month at home. Maximum duration is length of stay in the ICU plus 1 month at home.

SUMMARY:
The purpose of this project is to improve mobility in the perioperative period using activity trackers to augment current practice.

Delirium and poor functional status following ICU stays are intractable problems for which clear solutions do not exist. Digital health approaches have not been applied to these problems in the ICU setting and may represent a viable and unexplored intervention.

The program will involve the utilization of an activity tracker in ambulating patients. There will be two arms to the program. The first will involve the longitudinal study of ambulating lung transplant patients. Patients will be given an activity tracker at time of transplant which will continue throughout their care into their first month at home. The data will be collected to identify correlation between activity and clinical outcomes.

DETAILED DESCRIPTION:
Early mobilization of patients, minimizing sedatives, maximizing pain control, optimizing sleep are strongly associated with decreased rates of delirium, decreased ICU length of stay, decreased hospital length of stay as well as improved functional status and quality of life at 1 year. Cardiac surgical patients that are at high risk of prolonged stay in the ICU due to the inherent nature of their disease (ie need for MCS (mechanical circulatory support) or lung transplantation) are most likely to benefit from a systematic aggressive approach to early mobilization. Technology such as activity trackers and virtual reality have been studied in general surgical populations but with limited data in the ICU and to date no studies in a cardiac surgical population. Activity trackers utilized in a multidisciplinary team to provide objective data to care teams and patients can be used to develop goal setting and patient motivation for teams, thereby improving mobility

Overall Goal: To evaluate whether quantitative information on post procedural ambulation in mechanical device patients, cardiac surgical patients and lung transplant patients can improve care teams ability to monitor and identify patients at high risk for complications and prolonged length of stay.

* The purpose of the research is to improve mobility in the perioperative period using Activity Trackers to augment current practice.
* Objective quantification and improvement in activity of post cardiac surgery patients might result in improved clinical outcomes, thereby making this tool a part of routine practice.

Patient Populations:

1. Lung transplant patients
2. Routine postoperative Cardiac surgical patients (elective cardiac surgical procedures including CABG and Valve replacement)
3. Device Patients (axillary patients pre-open heart transplantation (OHT). Post MCS patients)

Specific Aim 1: Create standardized trajectories for ambulation of study subject populations from time of index procedure to 30 days postoperatively Specific Aim 2: To determine if deviation from the standardized trajectory of postoperative ambulation predicts disposition (home, rehabilitation facility or SNF), length of stay, 30 day readmissions, intensive care unit (ICU) readmission, DVT, respiratory insufficiency (aspiration) Specific Aim 3: To determine if decline in ambulation over 48 hours for a given patient predicts outcomes including length of stay, readmission to an icu, readmission to hospital, deep vein thrombosis (DVT), respiratory insufficiency.

The purpose of this project is to improve mobility in the perioperative period using activity trackers to augment current practice.

Delirium and poor functional status following ICU stays are intractable problems for which clear solutions do not exist. Digital health approaches have not been applied to these problems in the ICU setting and may represent a viable and unexplored intervention.

The program will involve the utilization of an activity tracker in ambulating patients. There will be two arms to the program. The first will involve the longitudinal study of ambulating lung transplant patients. Patients will be given an activity tracker at time of transplant which will continue throughout their care into their first month at home. The data will be collected to identify correlation between activity and clinical outcomes.

The second part of the program will be within the intensive care unit. The daily step count will be recorded for all ambulatory patients that fall into one of the defined subject populations and have signed informed consent. Step counts will be displayed for the care teams as well as the patient. This will be utilized by team to continuously evaluate and modify physical mobility goals for the patient with earlier recognition of decreasing mobility which is associated with worse outcomes. The goals and progress for the patient will be displayed to the nursing staff and the patient which we hypothesize will increase motivation.

Our hypothesis is that these interventions will increase mobility, decrease ICU length of stay, optimize the ICU experience, and potentially increase in 6-month functional status.

ELIGIBILITY:
Inclusion Criteria:

Patients that are at high-risk patients for one of the following interventions, will be considered for this study:

1. Axillary impella patients awaiting transplant, advanced MCS therapy or weaning
2. MCS patients post procedure including TAH, LVADs
3. Lung Transplant patients
4. Subjects > 18 years of age.
5. Ability to provide informed consent and follow-up with protocol procedures

Exclusion Criteria:

1. Non-ambulatory patients
2. Participation in an on-going protocol studying an experimental drug or device
3. Use of a walker, cane or wheelchair at baseline
4. Inability to wear the biosensor on the wrist
5. Any condition or other reason that, in the opinion of the Investigator or Medical Monitor, would render the subject unsuitable for the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Investigators and co-investigators will approach eligible subjects about the study in person after identification of patients in the intensive care unit or prior to surgery if it is not an emergent surgery. Some of the patients will be patients of other surgeons and intensivists who are part of the team-based care of these cardiac surgical patients.
Sampling Method: Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Daily ambulation | From date of inclusion until discharge from hospital assessed up to 30 days post enrollment
  Steps taken
Length of Stay | From date of inclusion until discharge from hospital assessed up to 30 days post enrollment
  Days until Discharge to a transitional care facility vs. home
Admit again to ICU | From date of inclusion until event or 30 days post enrollment
  Readmissions to an ICU or hospital

CONTACTS AND LOCATIONS:
Overall Officials: Anahat Dhillon, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States